CLINICAL TRIAL: NCT04092569
Title: The Effectiveness of Pre-medical Consultation (PMC) Diabetes Self-care Education Programme on Glycemic Control in Adults With Type 2 Diabetes
Brief Title: Effectiveness of Pre-medical Consultation Diabetes Self-care Education Programme on Glycemic Control in Type 2 Diabetes
Acronym: PMC-SEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, LAU Siu Wai Maggie, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019.255
Record Dates: First submitted 2019-08-06; First posted 2019-09-17 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Type 2 Diabetes
Keywords: Pre-medical Consultation self-care education; Glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: All patients who are 'newly referred for advanced diabetes management' from general practitioners or general out-patient clinic to specialist out-patient clinic of Alice Ho Miu Ling Nethersole Hospital from 1/8/2019 to 31/12/2019 will be recruited.
  After signing written informed consent on day of diabetes complication screening, they will be randomized into CG (n=10 for pilot study; n=60 for main study) or IG (n=10 for pilot study; n=60 for main study) groups, using sealed envelope, opened by an independent staff, containing randomly generated computer codes for group assignment. All patients will undergo diabetes complication screening including examination of eye and feet, collection of blood and urine samples and filling in DM questionnaires at baseline, and HbA1c with diabetes self-care questionnaires at 24 weeks (for IG only) and 36 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Pre-medical consultation structured diabetes self-care education programme
  Interventions: Behavioral: Pre-medical consultation structured diabetes self-care education programme
- Control group (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Pre-medical consultation structured diabetes self-care education programme — The findings of integrative review revealed positive effects of DSME in improving glycemic control and promoting self-care among people with type 2 diabetes.
  An evidence-based protocol is developed based on these findings to generate a DSME program for newly referred patients to SOPCs and before their first medical consultation to improve glycemic control and enhance self-care of people with type 2 diabetes in Hong Kong. The investigator will ensure that this study is conducted in compliance with ICH-GCP and in compliance with the Declaration of Helsinki.
  Arms: Intervention group

SUMMARY:
This proposed project is a prospective randomized controlled trial to examine the clinical effects of pre-medical consultation structured diabetes self-care education program on intervention group (IG) versus control group (CG) for patients with type 2 diabetes in a specialist outpatient clinic of a regional hospital.

DETAILED DESCRIPTION:
Protocol Revised Date: 23 April 2019

Introduction Diabetes Mellitus (DM) is known as one of the major causes leading to cardiovascular diseases, stroke, diabetes kidney diseases, blindness or non-traumatic lower limb amputations. It is estimated that one in ten people to have diabetes and it has been projected that one in three adults will develop type 2 diabetes by 2050. Similarly, the prevalence of Type 2 Diabetes Mellitus (T2DM) in Hong Kong is estimated to be one in ten in adult population.

DM is a progressive metabolic disease and necessitates continuous medical care, diabetes self-management education and skills training to prevent or delay development of acute and chronic complications. Educating patients with diabetes in self blood glucose monitoring, healthy eating, regular physical activities, medication adherence, stress management and smoking cessation are important behavioral modifications required in diabetes self-care education. Besides providing education, diabetes nurses provide support and discuss with patients regarding their concerns and worries about diabetes and empower them to live their life positively with diabetes.

The Service Gap

Patients with diabetes with or without cardiovascular or renal comorbidities, are inevitably a burden to healthcare system. In Hong Kong and most other countries, if not all, patients are referred to specialist out-patient clinics (SOPC) for more advanced diabetes management from either general out-patient clinics (GOPC) or private practitioners (GP). Hence, these new case referrals from GOPC or GP are patients already have established DM on oral anti-diabetic drugs and/or insulin injections and with diabetes complications. Nevertheless, they have to wait for a long period of time, approximately one to two years before they could be seen at SOPC.

The role of a diabetes nurse is recognized as providing diabetes education, individualized care, self-care promotion, teaching physical skills and enhancing psychological support. However, majority of DM patients are being first seen at general medical clinics, and only a proportion of them will be referred by case medical practitioner to diabetes nurses for education. In other words, the role of the diabetes nurses is quite 'passive' and the basic education program may fail to cover all newly referred patients.

According to Hospital Authority (HA) report, the waiting time for stable case new case booking in medicine specialist out-patient clinics from October 1, 2017 to September 30, 2018 is the median 94 weeks (= 24 months = 2 years) to the longest 119 weeks (= 30 months = 2.5 years) for first time medical consultation at SOPC. Most of them are with suboptimal glycemic control and/or co-morbidities, such as retinopathy or renal impairment at time of referral made and necessitate earlier medical management. Burden of diabetes on public health care system in Hong Kong is alarming. The number of patients with diabetes increased over 9,000 (31.5%) in five years from 2010 to 2015, with around 200,000 admissions for diabetes-related complications, which accounts for 18% of all admissions and around one million SOPC visits, which accounts for 14% of all SOPC attendance.

Thus, the clinical triggers are:

1. What is the impact of delivering pre-medical consultation nursing intervention or diabetes education to these newly referred patients with type 2 diabetes at SOPC?
2. What are the effects of early nursing consultation and diabetes self-care education on glycemic control and self-care in patients with type 2 diabetes?

Hypothesis Pre-medical consultation structured diabetes self-care education programme can provide significantly greater improvements in glycemic control and self-care behaviors in adults with type 2 diabetes than usual care.

Objectives

1. To evaluate the effectiveness of pre-medical consultation structured diabetes self-care education programme on glycemic control in adults with type 2 diabetes.
2. To assess the effectiveness of pre-medical consultation structured diabetes self-care education programme on diabetes-specific self-care behaviors.
3. To examine acceptability and usefulness of the intervention protocol by conducting a focus group interview on the intervention group.

Proposed evidence-based intervention protocol The findings of integrative review revealed positive effects of diabetes education in improving glycemic control and promoting self-care among adults with type 2 diabetes. An evidence-based protocol is developed based on these findings to generate a structured diabetes self-care education programme for newly referred patients before their first medical consultation at SOPC to improve glycemic control and enhance self-care in adults with type 2 diabetes in Hong Kong.

Study design This will be a randomized controlled trial to examine the effects and acceptability of a structured diabetes self-care education programme for type 2 diabetes patients as an intervention group (IG) versus a control group (CG) of usual care in a specialist out-patient clinic of a regional hospital.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes, age above 18 years old, who are 'newly referred' (established as well as newly diagnosed of DM) to specialist out-patient clinic at Alice Ho Miu Ling Nethersole Hospital
* Suboptimal glycemic control of glycosylated haemoglobin, HbA1c >7%
* Chinese and literate, able to answer questionnaires

Exclusion Criteria:

* Inability to give informed consent.
* Poor glycemic control with glycosylated haemoglobin, HbA1c >12% and/or related complications will receive early medical appointment or require hospital admission.
* Having advanced diabetes related complications, e.g. diabetes kidney disease with glomerular filtration rate (eGFR) <30 mL/min/1.72m2
* Life threatening condition with reduced life expectancy such as patients with cancer at terminal stage.
* Those with active mental disorders and learning disability.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Blood Glycosylated haemoglobin, HbA1c at 6 months | At baseline, week 24.
  Blood HbA1c will be taken at baseline diabetes complication screening, week 24 for both IG and CG.
Change from Baseline Blood Glycosylated haemoglobin, HbA1c at 9 months | At baseline, week 36.
  Blood HbA1c will be taken at baseline diabetes complication screening week 36 for both IG and CG.

SECONDARY OUTCOMES:
The Chinese version of the Diabetes Management Self-Efficacy Scale Questionnaire | At baseline, week 24 and week 36.
  The Diabetes Management Self-Efficacy Scale Questionnaire (C-DMSES) is a 20-item scale that assesses diabetes self-care, including blood glucose monitoring, dietary adherence and physical activity adherence. Participants are asked to read each of the 20 items and rate on a 0-10 Likert scale. Higher scale scores indicate better self-care behavior. This scale has been validated and shown satisfactory reliability (r=0.86) in research.
The Chinese version of the Diabetes Empowerment Scale Questionnaire - Short Form | At baseline, week 24 and week 36.
  The Chinese version of the Diabetes Empowerment Scale Questionnaire (C-DES) is a 10-item scale and includes five subscales: overcoming barriers, achieving goals, coping, determining suitable methods and obtaining support. Participants are asked to rate each of the 10 items on a 0-5 Likert scale. Higher scale scores indicate better self-efficacy. This scale has been validated and shown satisfactory reliability (r=0.95) in study.

CONTACTS AND LOCATIONS:
Overall Officials: Siu Wai Maggie LAU, MPhil, Principal Investigator — Chinese Univeristy of Hong Kong
Locations (1):
- Diabetes Centre, Alice Ho Miu Ling Nethersole Hospital, Tai Po, New Territories, Hong Kong